CLINICAL TRIAL: NCT05474365
Title: Stepwise Training Program: a Novel Practice Model for Laparoscopic Suturing
Brief Title: Stepwise Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: IRCAD-Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SHHstepwise01
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Laparoscopic Suturing
Keywords: laparoscopic suturing; stepwise training; practice schedule; laparoscopic skill acquisition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medical students (Experimental)
  Interventions: Other: Stepwise training
- Surgical trainees (Experimental)
  Interventions: Other: Stepwise training
- Attending Surgeons (No Intervention)

INTERVENTIONS:
Other: Stepwise training — The protocol of stepwise training is mentioned in Detailed description in Study Description.
  Arms: Medical students; Surgical trainees

SUMMARY:
Laparoscopic skills training is essential and has been correlated with intraoperative performance. There are a number of training curricula developed to shorten the laparoscopic learning curve. Laparoscopic suturing is an advanced technique of laparoscopic skills that requires high level of hand-eye coordination.

After obtaining basic laparoscopic skills, the trainees traditionally progress to learn intracorporeal suturing by serially repeating the multiple steps required to complete laparoscopic suture. It has been advocated that teaching of complex laparoscopic task should be divided into necessary steps. Therefore, the steps of intracorporeal suturing can be broken down into discrete blocks, such as needle pick up, passing needle, and forming a knot. The learner is to repetitively practice one step in one block to master the required skill before moving on to the next block. This form of blocked practice has been recognized effective and efficient for motor skill acquisition.

We established stepwise training program for laparoscopic intracorporeal suturing based on the concept of blocked practice for the medical students and surgical trainees in our institution. It is our hypothesis that the stepwise program will improve laparoscopic suturing techniques of the participants. The purpose of this study is to assess the learning outcomes of laparoscopic suturing learning outcomes after our novel stepwise training program.

DETAILED DESCRIPTION:
1. Application for Institution Review Board approval.
2. Voluntary participants were recruited from 5th-graded medical students, surgical trainees, and attending surgeons in single institution. An informed consent was obtained from the participants. The training courses and tests for medical students, surgical trainees and attending surgeons were described as follows:

   The medical students watched a pre-course video of laparoscopic suturing, followed by two 2-hour courses of stepwise training for laparoscopic suturing. A test of the standard laparoscopic suturing task was performed immediately after each course.

   The surgical trainees took single 2-hour course of stepwise training without watching the pre-course video. A test of the standard laparoscopic suturing task was performed before and after the course.

   Attending surgeons were invited to take the test as controls without joining the course.
3. Equipment and laparoscopic task The training and task were performed on iSuture laparoscopic training desk. A 3-0 polysorbTM (Covidien, GL-182) with a 20-cm length of thread was used for the laparoscopic task. The participants were required to fulfill an intracorporeal suture with a first double-throw knot, followed by two single-throw knots on the suture pad.
4. Stepwise training program

The instructor described the schedule to the participants in the beginning of the program. Two participants shared a set of the equipment and practiced in turn in blocks. At the beginning of each block, the step was demonstrated with video clips. The participants only practiced the specified step in the block before proceeding to the next block. The detailed schedule is listed as follows:

Pick up needle: 10 mins (5 mins for each hand) Control needle angle: 20 mins (10 mins for each participant) Needle drive and pull thread: 20 mins (10 mins for each participant) Make double throws: 20 mins (10 mins for each participant) Knot tying: 20 mins (10 mins for each participant) Free practice: 30 mins (15 mins for each participant)

ELIGIBILITY:
Inclusion Criteria:

* 5th-graded medical students
* Surgical trainees

Exclusion Criteria:

* did not consent for the data collection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
laparoscopic suturing competency assessment tool | 6 months
  All the tests were video recorded. The videos were processed with de-identification and random coding, and then reviewed independently by two expert surgeons (HC & CW) who were blinded to the identity of the test-taker. A previously validated tool, laparoscopic suturing competency assessment tool (LS-CAT), was used to evaluate the videos. LS-CAT is composed of four domains, "pick up needle", "pass needle through edges", "create first double wind", and "knot tying". A low score in LS-CAT represented a high level of skill set with a score of 8 indicating the best performance. Suturing time was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Hung Wei, MD, Study Director — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCluney AL, Vassiliou MC, Kaneva PA, Cao J, Stanbridge DD, Feldman LS, Fried GM. FLS simulator performance predicts intraoperative laparoscopic skill. Surg Endosc. 2007 Nov;21(11):1991-5. doi: 10.1007/s00464-007-9451-1. PMID 17593434
- [Result] Stefanidis D, Hope WW, Korndorffer JR Jr, Markley S, Scott DJ. Initial laparoscopic basic skills training shortens the learning curve of laparoscopic suturing and is cost-effective. J Am Coll Surg. 2010 Apr;210(4):436-40. doi: 10.1016/j.jamcollsurg.2009.12.015. PMID 20347735
- [Result] Thinggaard E, Bjerrum F, Strandbygaard J, Gogenur I, Konge L. Validity of a cross-specialty test in basic laparoscopic techniques (TABLT). Br J Surg. 2015 Aug;102(9):1106-13. doi: 10.1002/bjs.9857. Epub 2015 Jun 11. PMID 26095788
- [Result] IJgosse WM, Leijte E, Ganni S, Luursema JM, Francis NK, Jakimowicz JJ, Botden SMBI. Competency assessment tool for laparoscopic suturing: development and reliability evaluation. Surg Endosc. 2020 Jul;34(7):2947-2953. doi: 10.1007/s00464-019-07077-2. Epub 2019 Aug 26. PMID 31451918